### MCC-16-12518 NCT04468230

Phase 2 Study of Nicotine for the Treatment of Pain Associated with Chemotherapy-Induced Peripheral Neuropathy
10/21/2022

### RESEARCH PARTICIPANT CONSENT FORM

**TITLE:** Phase 2 Study of Nicotine for the Treatment of Pain Associated with

Chemotherapy-Induced Peripheral Neuropathy

**PROTOCOL #**: MCC-16-12518

**VCU IRB #:** HM20019616

**SPONSOR:** VCU Massey Cancer Center

**INVESTIGATOR:** Renato Martins, MD

VCU Massey Cancer Center 1201 East Marshall Street

Box 980070

Richmond, VA 23298

804-628-3121

### INTRODUCTION

This consent form will tell you about this research study, which is also called a clinical trial. Your study doctor or study team will explain the research study to you. Research studies only include people who choose to take part. You have the option to not participate. You may take home an unsigned copy of this consent form so that you can discuss the study with your family or friends before making your decision. You may also discuss it with your health care team. If you have any questions, ask your study doctor or study team for more explanation. Please take your time to make your decision about taking part in this study.

### **OVERVIEW AND KEY INFORMATION**

### Taking part in this study is your choice

You can choose to take part or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

### Why is this study being done?

Some of the chemotherapy and other drugs used to treat cancer can damage nerves that are around the body and outside of the brain and spinal cord (i.e., peripheral nerves). Peripheral nerves carry sensations (feelings) to the brain and control the movement of our arms and legs. They also control the bladder and bowel. When this happens, it is called chemotherapy-induced peripheral neuropathy (CIPN), a set of symptoms that include pain, burning, tingling, weakness, and loss of feeling or numbness. These symptoms may start in the hands and feet and may move to other parts of the body. CIPN can cause severe pain and can make it difficult to do things like walk, write, or button your shirt. If it gets very bad, it can cause more serious problems like changes in your heart rate and blood pressure, dangerous falls, trouble breathing, or loss of muscle function.

The purpose of this study is to test whether nicotine, in the form of a nicotine patch that is placed on the skin, can lessen the symptoms of CIPN. Another purpose of this study is to test 2 different doses of the nicotine patch and if see one dose works better than the other.

Up to 52 people will take part in this study.

### What is the usual approach to treating my CIPN

You are being asked to take part in this study because you have been diagnosed with CIPN. People who are not in a research study may be treated with other drugs or other treatments available for CIPN.

### What are my other choices if I do not take part in this study?

If you decide not to take part in this study, you have other choices. For example:

- You may choose to have duloxetine, tricyclic antidepressants, gabapentin, and topical applications (e.g., baclofen and ketamine) or another type of treatment, if any are available
- You may choose to take part in a different study, if one is available
- Or you may choose not to be treated for CIPN

### How will my CIPN be treated if I take part in this study?

This study will not change how your cancer is treated.

During the first treatment part of the study, you will place a nicotine patch that has a dose of 7 mg of nicotine on your arm every day for 14 days. You will need to keep your patch on for at least 16 hours per day. After 14 days, you will have a washout period of at least 14 days and possibly up to 21 days, which means you will not wear a nicotine patch during this time. Next, you will place a nicotine patch that has a dose of 14 mg of nicotine on your arm every day for 14 days for at least 16 hours per day.

During the 14 days that you are wearing the 7 mg and the 14 mg nicotine patch, you will be asked to visit the clinic about once a week. You will also be asked to visit the clinic at least once after you have finished using the nicotine patches.

You will be given a study drug diary and will be asked to write down when you put your nicotine patch on and when you take the nicotine patch off every day.

### How long will I be in this study?

If you do not have any serious side effects, you will be in this study for about 18 weeks or a little over 4 months.

After your last day of placing the 14 mg nicotine patch on your arm, your study doctor will continue to watch you for side effects and follow your condition for about 1 month or 30 days.

About 3 months after your last day of placing the 14 mg nicotine patch on your arm, your study doctor or research nurse will call you to see if you have continued using the nicotine patch to lessen your CIPN symptoms, and to ask you if you have developed a dependence or addiction to nicotine or products containing nicotine.

### What test and procedures will I have if I take part in this study?

If you decide to take part in this study, some of the exams, tests, and procedures you will have are part of the usual approach when treating your CIPN. Your study doctor or study team will tell you about these. The results of the usual exams, tests, and procedures may also be used for the research purposes of this study.

In addition to the regular exams, tests, and procedures, you will need to have blood tests to find out if you can take part in the study.

You will be asked to fill out some surveys with questions about your CIPN symptoms and how you feel. Researchers will use this information to learn more about how the nicotine patch affects CIPN symptoms. Each survey should take about 2 to 5 minutes. You don't have to answer any question that makes you feel uncomfortable.

You will also be asked to give one blood sample at each visit (about half of 1 teaspoon) that will be used to measure the amount of nicotine in your blood. This study will not use your samples to sequence all or part of your DNA. Blood samples remaining after the tests are completed will be destroyed.

You will be asked to fill out the surveys and give a blood sample during clinic visits at the following times during the study:

- Before beginning the study
- Week 2 of your 7 mg nicotine patch treatment
- Week 1 of your 14 mg nicotine patch treatment
- Week 2 of your 14 mg nicotine patch treatment
- During your 30-day follow-up period

Individual results of the research using your samples will not be provided to you, and there will be no benefit to you. The samples are collected only for this research study. If any inventions or discoveries result from the use of your samples, there are no plans to share any money or profits with you.

### What are the risks and benefits of taking part in this study?

### Risks

We want you to know about a few key risks right now. We give you more information in the "WHAT POSSIBLE RISKS CAN I EXPECT FROM TAKING PART IN THIS STUDY" section of this consent form.

Some of the most common side effects that the study doctors know about are:

- Dizziness
- Nausea
- Headache
- Mild itching or redness near the area that your nicotine patch is placed

There is a small risk that you could become addicted to or dependent on nicotine while using nicotine patches.

Participation in research might involve some loss of privacy.

### **Benefits**

There is no guarantee that you will receive any medical benefits from being in this study. The study drugs may or may not be make your CIPN symptoms better. Patients in the future may benefit from the knowledge gained through your participation in the study.

### WHAT POSSIBLE RISKS CAN I EXPECT FROM TAKING PART IN THIS STUDY?

You will be receiving nicotine through a patch that will be placed on your skin if you choose to take part in this study. There is a risk that the nicotine patch may not be as good as other drugs at treating your CIPN. There is also a risk that you could have side effects from the nicotine patch. These side effects may be worse and may be different than you would get with the usual approach for your CIPN.

The lists below are the most common and the most serious side effects that we know about. If important new side effects are found, your study doctor will discuss these with you. Here are important points about side effects:

- Your study doctor does not know who will or will not have side effects
- Some side effects may go away soon, some may last a long time, or some may never go away
- Some side effects may be serious and may even result in death

Here are important points about how you and your study doctor can make side effects less of a problem:

- Tell your study doctor if you notice or feel anything different so they can see if you are having a side effect
- Your study doctor may be able to treat some side effects
- Your study doctor may adjust the study drugs to try to reduce side effects
- Let your study doctor know of any questions you have about possible side effects. You can ask your study doctor questions about side effects at any time.

Common side effects associated with nicotine include:

- Dizziness
- Headache
- Nausea
- Skin Irritation
- Rapid heartbeat

Some less common side effects associated with nicotine include:

- Constipation
- Drowsiness
- Stomach cramps

Some rare side effects of nicotine include:

- Hives
- Seizures
- Irregular heart beat or palpitations
- Trouble breathing

We will watch you and other patients in this study very closely for any serious problems that could happen with a nicotine overdose and will mean that you need to stop using the nicotine patch:

- Severe headache
- Chest pain
- Irregular heartbeat or palpitations
- Swelling in the hands, ankles, and/or feet

The nicotine will be given to you in the form of a skin patch. Side effects that may occur near the area that your nicotine patch is placed include:

- Mild itching
- Redness
- Burning
- Stinging

### **Risk of Developing Nicotine Dependence**

There is a small risk that you could become addicted to or dependent on nicotine while using nicotine patches. There is a small risk that you will experience nicotine withdrawal side effects during the weeks that you are not using a nicotine patch (washout period) and after you remove the 14 mg nicotine patch on the last day of study treatment. Nicotine withdrawal side effects may occur within 4 to 24 hours after the removal of the nicotine patch and may last up to 3 days.

Common side effects associated with nicotine withdrawal include:

- Feelings of sadness or depression
- Headache
- Increased appetite
- Irritability
- Nausea
- Trouble sleeping

### **Risks Associated with Collection of Blood Samples**

Common side effects of blood sample collection are brief pain and bleeding or bruising at the puncture site used to collect the blood sample. There is also a small risk of infection, light-headedness, and fainting.

### Reproductive Risks

You should not get pregnant or breastfeed while taking part in this study. The effects of nicotine to an unborn child or breastfeeding child are not fully known.

If you are able to become pregnant, you will need to have a pregnancy test to find out if you can be in the study. If you participate in this study, you must agree to use a reliable method to prevent pregnancy during the study treatment. Check with the study doctor about what methods of preventing pregnancy are acceptable for you.

### Interactions with Other Medications, Supplements, and Food

There are numerous medications, herbal products, vitamins, and dietary products that can interact with the study drugs. Interactions with medications and supplements may cause more side effects or decrease the effectiveness of the study drugs or other medications. Your study team will review your current medications and supplements to be sure that there are no concerns before you start taking the study drugs. You should not start taking any new over-the-counter or prescription medications or supplements without first checking with your study team about possible interactions.

You will be given a pocket card that identifies this research study. Carry this with you at all times. You should show it to your health care providers so that they can check with your study doctor or study team member about possible interactions that may occur with new medications added while you are participating in this study.

### **Risk of Loss of Confidentiality**

Participation in research might involve some loss of privacy. Researchers will make every effort to protect your privacy, but there is a small risk that someone outside the research study could see and misuse information about you.

### **CAN I STOP TAKING PART IN THIS STUDY?**

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let the study doctor know as soon as possible so you can stop safely. If you stop, you can decide whether or not to let the study doctor continue to provide your medical information for the purpose of the study.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study. The study doctor may take you out of the study:

- If your health changes and the study is no longer in your best interest
- If you have serious side effects that require you to stop according to the rules of the study
- If new information becomes available
- If you do not follow the study rules; or
- If the study is stopped by the sponsor, the Food and Drug Administration (FDA), or the institutional review board (IRB), which is a group of people who review the research with the goal of protecting the people who take part in the study

If you withdraw from the study, data that has already been collected about you will remain part of the study database and may not be removed.

### WHAT ARE MY RIGHTS IN THIS STUDY?

Taking part in this study is your choice. No matter what decision you make, and even if your decision changes, there will be no penalty to you. You cannot lose medical care or any legal rights by agreeing to participate in this study.

### WHAT ARE THE COSTS OF TAKING PART IN THIS STUDY?

The nicotine patches will be supplied at no charge while you take part in this study.

You will not be charged for any costs related to the collection and testing of your blood for nicotine levels or surveys that are for research purposes. The blood samples and surveys are not used for testing that affects your care.

You and/or your health plan/insurance company will be billed for all standard costs of treating your CIPN, including the cost of tests, procedures, medicines, or hospital admissions to manage any side effects.

### WILL I BE PAID TO PARTICIPATE IN THE STUDY?

You will not be paid to take part in this study.

### WHAT HAPPENS IF I AM INJURED OR BECOME SICK BECAUSE I TOOK PART IN THIS STUDY?

If you are injured by, or become ill, from participating in this study, please contact your study doctor immediately. Medical treatment is available at the Virginia Commonwealth University Health System (VCU Health System). Your study doctor will arrange for short-term emergency care at the VCU Health System or for a referral if it is needed.

Fees for such treatment may be billed to you or to appropriate third party insurance. Your health insurance company may or may not pay for treatment of injuries or illness as a result of your participation in this study. To help avoid research-related injury or illness, it is very important to follow all study directions.

### WHO WILL SEE MY MEDICAL INFORMATION?

Your privacy is very important to us. The researchers will make every effort to protect it, but your information may be given out if required by law. However, the researchers will do their best to make sure that any information that is released will not identify you.

Your research information and your personal identifying information will be kept private through the use of password-protected electronic files, locked research areas, and study identification numbers. Blood samples obtained for research purposes will be stored with the same safeguards. The results of this research may be presented at meetings or in publications, but you will not be identified by name.

There are organizations that may inspect your records. These organizations are required to make sure your information is kept private, unless required by law to provide information. Some of these organizations are:

- Virginia Commonwealth University (VCU)
- VCU Institutional Review Board (IRB)
- Food and Drug Administration (FDA)
- National Cancer Institute (NCI)

In the future, the identifiers (like your name and birthday) could be removed from the information you provide for this study. After that removal, your information could be used for new studies without asking for your consent again. Those possible new studies could be done by this study team or other researchers.

### **USE AND DISCLOSURE OF PROTECTED HEALTH INFORMATION**

The Health Insurance Portability & Accountability Act (HIPAA) of 1996 provides for the protection of your health information from unauthorized use and disclosure. This section tells you what health information about you may be used and given out in the study and who may give and receive the information. By signing the consent form for this study, you agree that health information that identifies you may be used and disclosed as needed for this research.

### **Authority to Request Protected Health Information**

The following people and/or groups may request your protected health information:

- · Principal investigator and research staff
- Study sponsor
- Research collaborators
- VCU IRB
- Data and Safety Monitoring Committee
- · Government/health agencies
- · Others as required by law

### **Authority to Release Protected Health Information**

The VCU Health System (VCUHS) may release the information identified in this authorization from your medical records and provide this information to:

- Health care providers at the VCUHS
- · Principal investigator and research staff
- Study sponsor
- Research collaborators
- Data coordinators
- VCU IRB
- Data and Safety Monitoring Committee
- Government/health agencies
- · Others as required by law

Once your health information has been disclosed to anyone outside of this study, the information may no longer be protected under this authorization.

### Type of Information that may be Released

The following types of information may be used for the conduct of this research:

Complete health record

Diagnosis and treatment codes

Discharge summary

History and physical exam

Consultation reports

Progress notes

Laboratory test results

Information about HIV tests

Information about psychiatric care

### **Expiration of This Authorization**

This authorization will expire (end) when the research study is closed, or when there is no need to review, analyze, and consider the data generated by the research study, whichever is later.

### Right to Revoke Authorization and Re-disclosure

You may change your mind and revoke (take back) the right to use your protected health information at any time. Even if you revoke this authorization, the researchers may still use or disclose health information they have already collected about you for this study. If you revoke this authorization you may no longer be allowed to participate in the research study. To revoke this authorization, you must write to the investigator.

### WHERE CAN I GET MORE INFORMATION?

You may visit the NCI website at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

### WHO CAN ANSWER MY QUESTIONS ABOUT THIS STUDY?

The investigator and study staff named below are the best persons to contact if you have any questions or concerns about this study or to report side effects or injuries.

Renato Martins, MD VCU Massey Cancer Center 1201 East Marshall Street Box 980070 Richmond, VA 23298 804-628-3121

You can also contact a study team member at <a href="masseycpc@vcu.edu">masseycpc@vcu.edu</a> or the Evening/Weekend Doctor on Call at 804-828-0951; ask for the doctor carrying pager 9898.

The Office of Research can answer your general questions or concerns about your rights as a participant in this or any other research. Also, if you would like to speak to a person who does

not work directly with your study doctor and the study team or if you cannot reach your study doctor or a member of the study team, you may contact:

Virginia Commonwealth University Office of Research 800 East Leigh Street, Suite 3000 Box 980568 Richmond, VA 23298 804-827-2157 https://research.vcu.edu/human\_research/volunteers.htm

MCC-16-12518 Page 10 of 11 Version Date: 02/14/2023

### MY SIGNATURE AGREEING TO TAKE PART IN THIS STUDY

I have been given the opportunity to carefully read this consent form. All of the questions that I wish to raise concerning this study have been answered.

By signing this consent form, I have not given up any of my legal rights or benefits. My signature indicates that I freely consent to participate in this research study.

| Participant Name ( <i>Printed</i> ) | |
|---|---|
| Participant Name (Signature) | Date |
| Person Conducting Informed Consent Discussion ( <i>Printed Name</i> ) | |
| Person Conducting Informed Consent Discussion (Signature) | <br>Date |
| Signature of Investigator ( <i>If different than above</i> ) | <br>Date |